CLINICAL TRIAL: NCT02286726
Title: Phase II Study of CPX-351 (Cytarabine:Daunorubicin) Liposome Injection in Patients With Newly Diagnosed AML at High Risk for Induction Mortality
Brief Title: CPX-351 in Treating Patients With Newly Diagnosed, High-Risk Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0548; NCI-2014-02529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0548 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-10-31; First posted 2014-11-10 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (lower-dose (50 units/m^2) CPX-351) (Experimental): Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5 of a 28-day course. Patients with persistent disease may receive a second course with treatment on days 1 and 3.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Liposome-encapsulated Daunorubicin-Cytarabine
- Arm II (intermediate-dose (75 units/m^2) CPX-351) (Experimental): Patients receive intermediate-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Patients with persistent disease may receive a second course with treatment on days 1 and 3.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Liposome-encapsulated Daunorubicin-Cytarabine
- Arm III (standard-dose (100 units/m^2) CPX-351) (Experimental): Patients receive standard-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Patients with persistent disease may receive a second course with treatment on days 1 and 3.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase II trial studies the best dose and how well liposomal cytarabine-daunorubicin CPX-351 (CPX-351) works in treating patients with newly diagnosed acute myeloid leukemia and who are at risk for not responding well to treatment. Liposomal cytarabine-daunorubicin CPX-351 combines two chemotherapy drugs that are known to help each other work better, and may work to stop the growth of cancer cells by blocking the cells from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess preliminary efficacy (as determined by the rate of complete response [CR] or CR with incomplete blood count recovery [CRi]) of two or three dose levels of CPX-351 in patients with newly diagnosed acute myeloid leukemia (AML) at high risk for induction mortality, defined as 30-50% predicted risk of death by day 60, and to select the most promising dose level for further efficacy testing.

SECONDARY OBJECTIVE:

I. To confirm the rate of dose limiting toxicities, including induction mortality (at day 60) for two different sub-maximum tolerated dose (MTD) dose levels (50 and 75 U/m^2).

EXPLORATORY OBJECTIVES:

I. To investigate the effect of CPX-351 on immune response, as determined by the effect on recovery of functional pathogen-specific and leukemia-specific immune responses and the recovery and function of natural killer (NK) cells.

II. To investigate the role of troponin-T as an early marker for CPX-351-induced cardiotoxicity.

III. To investigate ex vivo the cytotoxicity of combination of Pim-1 proto-oncogene, serine/threonine kinase (Pim) kinase inhibitor(s) and CPX-351 on circulating leukemia cells.

OUTLINE:

INDUCTION: Patients are randomized to 1 of 2 arms. After safety is established for both dose levels, and escalation is deemed feasible, an additional arm will be studied at the standard dose level.

ARM I: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5 of a 28-day course. Patients with persistent disease may receive a second course with treatment on days 1 and 3.

ARM II: Patients receive intermediate-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Patients with persistent disease may receive a second course with treatment on days 1 and 3.

ARM III: Patients receive standard-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Patients with persistent disease may receive a second course with treatment on days 1 and 3.

CONSOLIDATION THERAPY: Patients achieving CR receive liposomal cytarabine-daunorubicin CPX-351 on days 1 and 3. Treatment may repeat every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for as long as the study doctor thinks it is needed, every 2-3 months for up to 1 year, and every 3-4 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily sign an informed consent form
* Pathological diagnosis of AML according to World Health Organization (WHO) criteria (with at least 20% blasts in the peripheral blood or bone marrow): newly diagnosed de novo AML; except for acute promyelocytic leukemia (APL); newly diagnosed secondary AML, defined as having a history of an antecedent hematologic disorder (myelodysplastic syndromes [MDS], myeloproliferative disease [MPD] or history of cytotoxic treatment for non-hematologic malignancy) or apparent de novo AML with MDS-associated karyotype
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Serum creatinine =< 2.0 mg/dL
* Serum total bilirubin =< 2.0 mg/dL
* Serum alanine aminotransferase < 3 times the upper limit of normal (ULN); Note: If elevated liver enzymes are related to disease alanine aminotransferase (ALT) should be < 5 times ULN
* To be considered at high risk for induction mortality patients must have 1 or 2 of the following risk factors (patients >= 60 must have at least 1 risk factor, patients < 60 must have at least 2 risk factors) present; at least one risk factor in every patient must be an AML-related factor:

  * AML-related factors include:

    * Antecedent hematologic disorder (AHD) (MDS, chronic myelomonocytic leukemia [CMML], or MPD) or history of exposure to cytotoxic chemotherapy [therapy-related (t)-AML]), or WHO-defined AML with MDS-related changes or apparent de novo AML with MDS-associated karyotype
    * Unfavorable cytogenetics as defined by the European Leukemia Net
  * Patient-related factors:

    * Age >= 70
    * ECOG performance status (PS) >= 2
  * Co-morbidities:

    * Serum creatinine > 1.3 g/dL
* Cardiac ejection fraction >= 50% by echocardiography or multi gated acquisition (MUGA) (when left ventricular ejection fraction [LVEF] expressed as a range, at least the upper limit should include 50%)
* Able to adhere to the study visit schedule and other protocol requirements
* All men and women must agree to practice effective contraception during the study period if not otherwise documented to be infertile

Exclusion Criteria:

* Patients with history of second malignancy are eligible if they have documentation of disease stability, off therapy, based on computed tomography (CT) scan or other measures for the 6 months prior to entry in core
* Any serious medical condition or psychiatric illness that would prevent the patient from providing informed consent
* Chemotherapy or other investigational anticancer therapeutic drugs in the two weeks prior to study entry; in the event of rapidly proliferative disease, however, the use of hydroxyurea is permitted up to 24 hours before study entry in core
* Evidence of active central nervous system (CNS) leukemia
* Pregnant or lactating women
* Uncontrolled infection; to be eligible, patients receiving treatment for an infection (antibiotic, antifungal or antiviral treatment) must be afebrile (< 38.3 degrees Celsius [C]) and without hemodynamic instability or dyspnea from pneumonia for > 48 hours (hrs) prior to the start of induction therapy
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-metabolism disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghayas Issa, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2015 to January 2020
Period: Overall Study
Arm/Group | Arm I (Lower-dose (50 Units/m^2) CPX-351) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) | Arm III (Standard-dose (100 Units/m^2) CPX-351)
Started | 16 | 24 | 16
Completed | 16 | 24 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lower-dose (50 Units/m^2) CPX-351) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) | Arm III (Standard-dose (100 Units/m^2) CPX-351) | Total
Number analyzed (Participants) | 16 | 24 | 16 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 5 | 22
  >=65 years | 8 | 15 | 11 | 34
Age, Continuous [Median (Full Range); unit: years] | 63 [54 to 80] | 66 [53 to 82] | 69 [60 to 80] | 67 [53 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 4 | 19
  Male | 9 | 16 | 12 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 14 | 24 | 16 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 24 | 16 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response is defined as Complete response (CR) or CR with incomplete blood count recovery (CRi) rate: Complete Remission (CR) is Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 10^9/L (1000/μL); platelet count >100 x 10^9/L (100,000/μL). Complete Response with incomplete blood count recovery (CRi) is All CR criteria except for residual neutropenia (<1.0 x 10^9/L [1000/μL]) and/or thrombocytopenia (<100 x 10^9/L [100,000/μL]).
Time Frame: Up to 8 weeks (after induction therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lower-dose (50 Units/m^2) CPX-351) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) | Arm III (Standard-dose (100 Units/m^2) CPX-351)
Number analyzed (Participants) | 16 | 24 | 16
Participants
  Complete Response (CR) | 3 | 6 | 7
  Complete Response with incomplete blood count recovery (CRi) | 0 | 3 | 0

2. Secondary Outcome: Number of Participants Who Experienced Dose-limiting Toxicity (DLT)
Description: Defined as induction mortality (death occurring on or before day 60), grade 3 or 4 non-hematologic toxicity, or dose limiting hematologic toxicity at least possibly related to the study drug occurring during the first 28 days from the start of therapy. Estimated for each arm with 95% confidence intervals. Fisher's exact test will be used to compare the toxicity rate between the two dose levels.
Time Frame: Up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lower-dose (50 Units/m^2) CPX-351) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) | Arm III (Standard-dose (100 Units/m^2) CPX-351)
Number analyzed (Participants) | 16 | 24 | 16
Participants | 5 | 3 | 3

ADVERSE EVENTS:
Time Frame: up to 4 years
Arm/Group | Arm I (Lower-dose (50 Units/m^2) CPX-351) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) | Arm III (Standard-dose (100 Units/m^2) CPX-351)
All-Cause Mortality (participants affected / at risk) | 6/16 | 3/24 | 4/16
Serious Adverse Events (participants affected / at risk) | 11/16 | 15/24 | 11/16
Other Adverse Events (participants affected / at risk) | 0/16 | 11/24 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lower-dose (50 Units/m^2) CPX-351) (N=16) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) (N=24) | Arm III (Standard-dose (100 Units/m^2) CPX-351) (N=16)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 6 (7) | 2 (2)
Fever (General disorders) | 3 (6) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infection Right Arm Abcess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (3) | 4 (4)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 4 (6) | 4 (5)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1) | 1 (1)
Orbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lower-dose (50 Units/m^2) CPX-351) (N=16) | Arm II (Intermediate-dose (75 Units/m^2) CPX-351) (N=24) | Arm III (Standard-dose (100 Units/m^2) CPX-351) (N=16)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase Increase (Investigations) | 0 (0) | 1 (1) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Blood Bilirubin Increase (Investigations) | 0 (0) | 1 (1) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Ejection Fraction Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gastric Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Investigation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 4 (4) | 4 (4)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Vascular Disorders (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT02286726/Prot_SAP_000.pdf